CLINICAL TRIAL: NCT03267342
Title: Financial and Mental Health: Exploratory Research
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1504015686; 5R34MH107633-02 (NIH)
Record Dates: First submitted 2017-08-28; First posted 2017-08-30 (Actual); Last update posted 2018-06-29 (Actual); Status verified 2018-06

CONDITIONS: Financial Difficulties

STUDY DESIGN:
Intervention Model Description: Investigators will be testing four main interventions for clients of a Community Mental Health Center (CMHC) with serious mental illnesses who currently have control of their finances, based on our study of the literature on financial health and our preliminary research at CMHC. Participating clients will be free to choose which of the services to access and will be free to withdraw at any time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All participants (Experimental): low-income people with mental illness will be given one-on-one financial counseling, a weekly peer support group, supported access to mainstream banking services and access to a matched savings account for a 12-14 month period.
  Interventions: Behavioral: One-on-one financial counseling; Behavioral: Peer support group; Behavioral: Supported access to mainstream banking services; Behavioral: A matched savings account

INTERVENTIONS:
Behavioral: One-on-one financial counseling — Clients will be given access to one-on-one financial counseling, provided by trained peer specialists, initially working under the guidance of the project director. The Consumer Financial Protection Bureau's Your Money, Your Goals: Financial Empowerment Toolkit for Social Services Programs (21) will be used as a reference during counseling sessions, with a view to developing a manual based on clients' existing experiences and coping strategies, such that the desired behavior change is manageable, realistic, and based on real-life possibilities rather than idealized circumstances which may be far from the reality of people's lives. Counseling will in all cases be responsive to clients' particular needs and concerns, rather than following a predetermined sequence.
Behavioral: Peer support group — Support groups, facilitated by peer specialists and guided initially by the project director, will be offered for clients interested in specific financial issues such as budgeting, managing benefits, wise spending, planning and saving. The peer support groups will focus on enabling clients to share their own experiences with finances.
Behavioral: Supported access to mainstream banking services — Interested clients will be helped to open bank accounts at banks of their choice, and to manage associated tools such as Automatic Teller Machine (ATM) cards and online bill pay. Clients will also be advised regarding use of non-bank financial products such as prepaid cards and check cashers. Representatives from both bank and non-bank providers will be invited to come in and talk with clients about the services they offer, and clients will also be invited to visit the facilities to be guided around the available services.
Behavioral: A matched savings account — Clients will have the option of joining a savings club, which will combine group meetings, facilitated by a peer specialist under the initial guidance of the project director, and regular savings deposits towards specified goals. Clients will be offered a limited savings match as an incentive to achieve their savings goal (for example, the savings club will offer a 50% match on any money saved within a specified time period towards a specific goal, up to a maximum of a $100 match).

SUMMARY:
This project will develop a model for providing low-income people with mental illness with supports that enable them to manage their money as well as possible so that they are better able to meet their basic needs, to experience less anxiety about finances, and to live fulfilling lives in the community with the greatest possible degree of independence. The project will work within a citizenship-oriented approach to mental health care, which promotes recovery through linking people with mental illness to the rights, responsibilities, roles, resources and relationships necessary to achieve full membership in society. The aims of the project are to: train clinicians and peer staff so that they are able to integrate discussion of financial issues and concerns into their work with clients; provide on-site services including financial counseling, peer support groups, help with opening a bank account, and a savings club, and; develop a 'financial health' model which can be replicated by other providers of mental health services. The investigators hypothesize that the intervention will result in improved financial health, reduced financial stress, increased community participation, and improved satisfaction with care.

DETAILED DESCRIPTION:
This study will pilot and assess financial health interventions that will provide clients with financial counseling, and information about and access to financial management tools within the framework of citizenship-oriented care, which approaches recovery by linking clients to the 5 Rs of rights, responsibilities, roles, resources and relationships needed to achieve full membership in society. Based on results of previous research, the investigators hypothesize that the intervention will result in improved financial health, reduced financial stress, increased community participation, and improved satisfaction with care for the target group.

ELIGIBILITY:
Inclusion Criteria:

* All participants will be adults (18 years or older).
* Participants will be clients receiving services from the CMHC.
* The investigators intend to include clients who do not have a representative payee and who are employed, or receiving supported employment services at CMHC, or interested in employment

Exclusion Criteria:

* factors that compromise an individual's ability to provide informed consent such as a co-occurring organic brain syndrome or dementia
* age under 18, as the mental health center serves adults only.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Financial health measure | up to 15 months
  Improved financial health, defined as being more financially secure, and better able to plan for the future. This outcome was measured through questions about having a bank account, savings behavior, borrowing behavior, debt, financial advice, lending behavior, credit score, knowledge about credit score, perception of financial well-being, and financial attitudes.

SECONDARY OUTCOMES:
Citizenship instrument | up to 15 months
  The citizenship measure is an instrument developed through community-based participatory and concept mapping methods including a co-researcher group of persons with mental illnesses. The measure has been validated as psychometrically sound, with the measure and its domains demonstrating good internal consistency and construct validity.
  The Citizenship instrument is a quantitative survey which with a score from 1-5 where a higher score indicates a higher level of citizenship.
Wellness in 8 Dimensions Inventory | up to 15 months
  A measure that outlines wellness strategies that people may use for their personal recovery. The wellness in 8 dimensions inventory is a quantitative survey with a score from 1-4 where a higher score indicates greater wellness.
Financial Stress | up to 15 months
  This outcome was measured through asking participants about their financial steps levels and their stress about debt in particular.
Satisfaction with CMHC Care | up to 15 months
  This outcome was measured through asking how satisfied a person was with the care they receive at the mental health center, and whether they would recommend it to others.
Money mismanagement Measures | up to 15 months
  Money mismanagement was measured quantitatively using the money mismanagement measure which includes five constructs, each scored between 0-4, with a higher score indicating worse money mismanagement (except for construct B) (note that constructs A and G were cut from the original measure):
  B: Responsible Spending (scored negatively) C: Perceived Problem Managing Money D: Victimization E: Impulsive spending F: Spending for Drugs and Alcohol

CONTACTS AND LOCATIONS:
Overall Officials: Michael Rowe, Principal Investigator — Yale University